CLINICAL TRIAL: NCT01602783
Title: Use of 11C Acetate Imaging for Improved Prediction of the Effectiveness of Salvage Pelvic Radiation Post Prostatectomy: A Pilot Study
Brief Title: 11C Acetate Imaging Post Prostatectomy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow accrual; no further funding
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Umar Mahmood, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 10-464
Record Dates: First submitted 2012-05-17; First posted 2012-05-21 (Estimated); Last update posted 2014-03-18 (Estimated); Status verified 2014-03

CONDITIONS: Prostate Cancer
Keywords: Radical Prostatectomy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 11C Acetate Imaging (Experimental): 11C acetate imaging
  Interventions: Other: 11C Acetate Imaging

INTERVENTIONS:
Other: 11C Acetate Imaging — Single scan

SUMMARY:
This research is being conducted to test an imaging technique that may be able to detect small amounts of prostate cancer that can not be detected by standard imaging.

Many patients who are diagnosed with prostate cancer undergo surgery to remove the prostate. After this surgery, some patients have a PSA blood test that reveals a low but detectable level of PSA. This PSA may be produced by cancer cells in one of two locations: (1) near the area where the prostate used to be, or (2) elsewhere in the body. If the cancer is only in the area where the prostate used to be, it can be successfully treated with radiation to that area. If the cancer is elsewhere, radiation is not helpful. Currently, there is no available scan that can detect cancer when the PSA is still so low.

The test used in this study is called [11C] acetate PET screening. [11C] acetate is a radioactive tracer that is given by vein to patients before PET scanning. The PET scanner then detects radioactivity from the tracer that is attached to cells within your body and uses this information to create images (pictures) on a computer screen.

[11C] acetate PET scanning has been shown in early studies to detect smaller amounts of prostate cancer that can be detected by standard imaging tests such as CT scan and bone scan. If it is successful at detecting very small amounts of prostate cancer, [11C] acetate PET scanning will help doctors identify patients who will benefit from radiation therapy after their prostate has been surgically removed. It will also help them identify patients who have small amounts of prostate cancer in other parts of the body and will not benefit from radiation to the prostate area.

This type of PET scan is investigational. "Investigational" means that the scan is still being studied and that research doctors are trying to find out more about it. It also means that the FDA has not approved this type of PET scan for your type of cancer. The information collected by this scan will determine whether this type of scanning is helpful but it will not be used to make decisions about your medical care.

DETAILED DESCRIPTION:
If you decide to participate in the study and are eligible, you will undergo a single [11C] acetate PET scan. This scan is designed to detect small amounts of your tumor that were not detected by the CT scan or the bone scan. On the day of the scan, you will fast for at least four hours prior to being given the tracer injection by vein. You will then be scanned in the PET scanner. The entire procedure will take approximately 2 hours.

The investigators would like to keep track of your medical condition after you have completed your scan. The investigators would like to do this by looking up information in your medical record during the year following the scan to see how you are doing. Checking your condition helps us understand whether the [11C] acetate PET scan will be helpful to other patients in the future.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the prostate
* History of radical prostatectomy
* Age ≥18 years
* PSA ≥0.5 and <4.0 ng/mL
* Abdominal-Pelvic CT scan without evidence of prostate cancer
* 99mTc MDP bone scan without evidence of prostate cancer
* Patient and clinician decision to proceed to salvage pelvic radiation therapy

Exclusion Criteria:

* Presence of known extra-pelvic evidence of prostate cancer
* Unable to fast for 4 hours
* Uncontrolled diabetes
* History of bilateral orchiectomies
* Ongoing treatment with any systemic therapy intended for the treatment of prostate cancer

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2011-12; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Sensitivity of 11C Acetate PET | 1 year
  Preliminarily demonstrate that the 11C acetate PET imaging of subjects who have experienced PSA relapse after prostatectomy for prostate cancer is more sensitive than currently available imaging techniques. Enrolled participants will have no evidence of recurrent disease on gold-standard imaging with CT abdomen/pelvis and 99mTc MDP bone scan (approximate sensitivity of 0%). The primary outcome is evidence of residual/recurrent disease as demonstrated by 11C acetate PET uptake outside of the prostatectomy bed.

SECONDARY OUTCOMES:
Establish a Preliminary Institutional Experience with 11C Acetate Imaging | 1 year
  To establish a preliminary institutional experience with 11C acetate imaging of men with prostate cancer
Correlate 11C Acetate PET Imaging Findings with PSA Evidence of Response | 1 year
  To descriptively correlate 11C acetate PET imaging findings with PSA evidence of response to subsequent salvage radiation therapy at 3 months and 6 months after the conclusion of radiation

CONTACTS AND LOCATIONS:
Overall Officials: Umar Mahmood, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States